CLINICAL TRIAL: NCT03619291
Title: Acute Effects of High-intensity Functional Circuit Training on Cognitive Function: a Randomised, Controlled Trial
Brief Title: High-intensity Functional Circuit Training and Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Prof, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SpM2018-001
Record Dates: First submitted 2018-07-27; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Exercise; Cognition
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity functional training (Experimental): all-out exercise
  Interventions: Other: High-intensity functional training
- Aerobic exercise (Active Comparator): walking
  Interventions: Other: Aerobic Exercise
- control (Sham Comparator): sitting
  Interventions: Other: control

INTERVENTIONS:
Other: Aerobic Exercise — walking on a treadmill at moderate intensity, total duration 15 minutes
  Arms: Aerobic exercise
Other: High-intensity functional training — functional exercises in circuit format at 20/10 s (work/rest) intervals, total duration 15 minutes
  Arms: High-intensity functional training
Other: control — physical inactivity, reading sports science literature, total duration 15 minutes
  Arms: control

SUMMARY:
The study investigates the acute effects of one bout of high-intensity functional circuit training on cognitive function against no-activity control and aerobic exercise.

DETAILED DESCRIPTION:
Exercise has been shown to acutely improve cognitive function (CF). However, it is unknown as to how high-intensity functional circuit training (HIFCT) affects CF. This study aims to compare the acute effects of one HIFCT bout against an inactive control condition as well as against one bout of conventional aerobic exercise.

Healthy participants will be randomly allocated to either a HIFCT group, an aerobic exercise group (walking) or an inactive control group. In the HIFCT group, participants perform a 15-minute workout, which is composed of functional exercise mimicking activities of daily living (e.g. squat, step-ups) and conducted in a circuit format. Each exercise is performed at all-out intensity for 20 seconds, followed by a 10-second break. Thus, the 15-min workout consists of 30 exercise intervals.

In the control group, participants will be inactively seated for 15 minutes, reading sports brochures and literature.

In the walking group, participants will walk at moderate intensity on a treadmill for 15 minutes.

Outcomes assessed pre and post-workout include the stroop test, trail making test, stop-signal task, heart rate, subjective arousal, rate of perceived exertion and exercise enjoyment.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years

Exclusion Criteria:

* severe orthopaedic, psychiatric, neurological, endocrine or cardiovascular disorders
* acute illness, not completely healed injuries
* muscle soreness
* pregnancy/nursing period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
interference control | 2 min
  stroop test

SECONDARY OUTCOMES:
cognitive flexibility/visual orientation | 2 min
  trail making test
inhibitory control | 2 min
  stop-signal task

IPD SHARING:
Plan to Share IPD: Undecided